CLINICAL TRIAL: NCT07365735
Title: A Prospective, Randomized, Controlled Trial of the TearCare MGX™ System With and Without Warming Hold (Xtend)
Brief Title: A Prospective, Randomized, Controlled Trial of the TearCare MGX™ System With and Without Warming Hold
Acronym: XTEND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN1 10280
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Meibomian Gland Dysfunction (Disorder)
Keywords: TearCare; XTEND; Meibomian Gland Dysfunction; MGD
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TearCare MGX with Warming Hold (Active Comparator): 15 minute thermal treatment with TearCare MGX followed by 10 minute warming hold
  Interventions: Device: localized heat therapy
- TearCare MGX without Warming Hold (Active Comparator): 15 minute thermal treatment with TearCare MGX without subsequent warming hold period
  Interventions: Device: localized heat therapy

INTERVENTIONS:
Device: localized heat therapy — Blink-assisted, open eye therapy. Heat (45 degrees C) applied for 15 minutes to the upper and lower eyelids, followed by manual expression of the meibomian glands.

SUMMARY:
TearCare is an office-based thermal therapeutic eyelid technology cleared by the US Food and Drug Administration for the treatment of evaporative dry eye disease due to meibomian gland dysfunction. In this randomized study, TearCare procedures using the TearCare MGX System (study device) with the extended Warming hold feature will be compared with TearCare procedures using the TearCare MGX System without the Warming hold (control group).

DETAILED DESCRIPTION:
This study will collect data to assess the clinical utility of the Warming Hold period. The TearCare MGX Warming hold is a 10-minute period beyond completion of the Core Therapy time that serves to preserve elevated temperature by outputting only enough energy to maintain heat at the lowest setting of the system. At the minimum warmth setting the SmartLid device surfaces provide a steady state temperature of 39.0°C.

This is a prospective, randomized, assessor-masked, single-center, non-significant risk (NSR) study. To reduce potential bias in the study, study staff performing the endpoint assessments will be masked. Subjects will also be masked as to group assignment.

In this randomized study, TearCare procedures using the TearCare MGX System (study device) with the extended Warming hold feature will be compared with TearCare procedures using the TearCare MGX System without the Warming hold (control group).

TearCare procedures in this study will include an in-office eyelid debridement, 15-minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects will receive one in-office TearCare procedure at the Procedure Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 22 years of age or older
2. Reports dry eye symptoms within the past 6 months
3. OSDI score of 23 to 79
4. Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤12 in each eye.
5. At least 15 glands in each lower eyelid should be expressible, with a sterile cotton swab, at the slit lamp.
6. Best corrected visual acuity of 20/100 or better, OU.
7. Willing and able to comply with the study procedures and follow-up
8. Understands and signs the informed consent.

Exclusion Criteria:

1. Use of:

   1. Cyclosporine, Xiidra, or serum tears within 60 days prior to Screening;
   2. Antihistamines (oral or topical) within 7 days prior to Screening;
   3. Oral tetracyclines or azithromycin within 30 days prior to Screening;
   4. Topical ophthalmic antibiotics, anti-glaucoma medications, steroids, non-steroidal anti-inflammatory medications within 30 days prior to Screening
   5. Isotretinoin (e.g. Accutane) at any time.
2. Any of the following dry eye treatments:

   1. Office-based dry eye treatment (e.g. IPL, TearCare, thermal pulsation [LipiFlow], iLux etc.) within 12 months prior to Screening either as part of routine care or clinical investigation;
   2. Planned or recent surgical procedures to the eye or eyelid (90 days prior to Screening);
   3. Meibomian gland expression within 6 months prior to Screening;
   4. Blephex or debridement within 3 months prior to Screening;
   5. Punctal occlusion (including collagen, e.g. Soft Plug, UltraPlug, or crosslinked hyaluronic acid, e.g. Lacrifill) or punctal plugs within 15 days of the Screening visit;
   6. Use of tear neurostimulators (i.e., True Tear, iTear100, Tyrvaya) within 2 weeks of the baseline visit. (Subjects must refrain from using tear neurostimulators for the duration of the study);
   7. Any history of meibomian gland probing.
3. History of eyelid, conjunctiva, or corneal surgery (including refractive surgery) within 12 months prior to Screening.
4. Any history of chalazion surgery, surgery on the tarsal conjunctiva, radial keratotomy (RK), complicated blepharoplasty, lid reconstruction, or significant complications post-refractive surgery.
5. Contact lens use within 2 weeks of the Procedure visit. Subjects presenting at the Screening visit using contact lenses must agree to discontinue use for a full 2 weeks (14 days) prior to the Procedure visit.
6. Active hordeolum, stye, or chalazion at the time of the Screening visit.
7. History of Herpes Simplex or Herpes Zoster of the eye or eyelid.
8. Any active, clinically significant ocular or peri-ocular infection, inflammation, or irritation.
9. Recurrent clinically significant eye inflammation, other than dry eye, within 3 months prior to Screening.
10. Clinically significant anterior blepharitis. In addition, collarettes or flakes of more than one quarter of the eyelid are excluded.
11. Clinically significant eyelid abnormalities in either eye (e.g. entropion/ectropion, blepharospasm, aponeurotic ptosis, lagophthalmos, distichiasis, trichiasis).
12. Clinically significant dermatologic or cutaneous disease of the eyelid or periocular area.
13. In the clinical judgement of the Investigator, meibomian glands have significant capping, atrophy, or are unable to be expressed, digitally or with a cotton swab.
14. Corneal surface abnormalities such as corneal epithelial defects (other than punctate staining), ulcers, corneal epithelial dystrophies, keratoconus, and ectatic disease of the cornea
15. Any active, clinically significant allergic, vernal, or giant papillary conjunctivitis.
16. Ocular trauma within 3 months prior to Screening.
17. Known history of diminished or abnormal facial, periocular, ocular or corneal sensation
18. Systemic diseases, in the Investigator's medical judgement, resulting in dry eye (e.g. autoimmune diseases such as Sjogren's syndrome, rheumatoid arthritis, lupus, Graves' disease, sarcoidosis, etc.)
19. Subject is currently using Retin A /Retin A derivatives.
20. Subject has permanent eyeliner/lid tattoos, eyelash extensions or wears false eyelashes.
21. Subject is currently using Latisse, Lash Boost or any other type of eyelash growth serum. Prostaglandin analog products such as Latisse should not be used within 30 days of the Screening visit.
22. Temporary false eyelashes, lash extensions, or any other type of false eyelash within 15 days of the Screening Visit.
23. Allergies to silicone tissue adhesives, acrylates and/or copper.
24. Subject has a pacemaker or implantable cardiac defibrillators (ICD).
25. Co-existing condition, either ocular or non-ocular that, in the judgement of the Investigator could affect the safety or effectiveness of treatment or the compliance of the subject to the protocol.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean difference between eyes in Meibomian Gland Secretion Score (MGSS) | MGSS used to calculate the difference in MGSS between eyes is obtained post-treatment at the procedure visit (Day 0).
  The Meibomian Gland Secretion Score (MGSS) grades the consistency of secretions from the meibomian glands. Fifteen meibomian glands in each of the lower eyelids were gently pressed and the secretions were scored on the scale below. Sum of the grade (0 - 3) for each of the 15 glands. Range for this score is 0-45. A higher number indicates more normal meibomian gland activity.
  Score Description of Secretion:
  0 - Nothing
  1. - Toothpaste
  2. - Cloudy
  3. - Clear The difference between eyes in the MGSS is the score for the right eye minus the score for the left eye. The mean is the arithmetic mean of this difference for all subjects.

SECONDARY OUTCOMES:
Mean change from Screening visit baseline in MGSS | MGSS is assessed at the Screening visit (Day -30 to Day -7) and at the Procedure visit (Day 0)
  The Meibomian Gland Secretion Score (MGSS) grades the consistency of secretions from the meibomian glands. Fifteen meibomian glands in each of the lower eyelids were gently pressed and the secretions were scored on the scale below. Sum of the grade (0 - 3) for each of the 15 glands. Range for this score is 0-45. A higher number indicates more normal meibomian gland activity. Score Description of Secretion: 0 - Nothing 1 - Toothpaste 2 - Cloudy 3 - Clear The change from baseline in the MGSS is the score obtained following treatment at the procedure visit minus the score obtained for the same eye at the Screening visit. The mean is the arithmetic mean of this difference for all eyes.
Mean change from Screening visit baseline in Meibomian Glands Yielding Any Liquid (MGYAL) | MGYAL is assessed at the Screening visit (Day -30 to -7) and at the Procedure visit (Day 0)
  The Meibomian glands yielding any liquid (MGYAL) is the number of glands in the lower eyelid secreting any liquid, (regardless of graded quality). The score can range from 0 (no glands secreting liquid), to 15 (all 15 glands with liquid secreted). A higher score is better. The mean change from Screening visit baseline is the mean difference between the MGYAL at screening and the MGYAL post-procedure at the procedure visit.
Mean change from Screening visit baseline in Meibomian Glands Yielding Clear Liquid (MGYCL) | MGYCL is assessed at the Screening visit (Day -30 to Day -7) and post-treatment at the Procedure visit (Day 0)
  The Meibomian glands yielding clear liquid (MGYCL) is the number of glands in the lower eyelid secreting clear liquid. The score can range from 0 (no glands secreting clear liquid), to 15 (all 15 glands with clear liquid secreted). A higher score is better. The mean change from Screening visit baseline is the mean difference between the MGYCL at screening and the MGYCL post-procedure at the procedure visit.
Subject Comfort during expression of second lid | Subject Comfort during expression of second lid is assessed post-treatment at the Procedure visit (Day 0)
  Subject Comfort during expression of second lid is assessed following treatment using a subject completed Likert scale rating the relative comfort of eyelid gland expression for the first lid expressed versus the second.
Ease of expression | Ease of expression is assessed following treatment at the Procedure visit (Day 0)
  Ease of expression is assessed following treatment using a masked-assessor completed Likert scale rating the relative ease of eyelid gland expression for the first lid expressed versus the second.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chester, OD, Principal Investigator — Cleveland Eye Clinic; Jaime Dickerson, PhD, Study Director — Sight Sciences, Inc.
Locations (1):
- Cleveland Eye Clinic, Brecksville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Protection of patient confidentiality.